CLINICAL TRIAL: NCT00475943
Title: Biomechanics of Human Epiglottal Movement and Inversion
Brief Title: Movement of Epiglottis During Swallowing
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 070156; 07-N-0156
Record Dates: First submitted 2007-05-18; First posted 2007-05-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-09-01

CONDITIONS: Deglutition; Dysphagia
Keywords: Swallowing Disorders; Swallowing; Videofluoroscopy; Dysphagia; Epiglottis; Healthy Volunteer; HV
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will examine how the airway closes during swallowing to prevent food or liquid from entering the voice box or lungs while eating or drinking. It will also test whether electrical stimulation of muscles in the neck can close the airway as it would close during swallowing. The long-term goal of this research is to determine the feasibility of a new approach for helping patients with a severe and life threatening swallowing disorder.

Healthy normal volunteers between 18 and 65 years of age who can swallow normally may be eligible for this study. Candidates are screened with a medical history, physical examination, electrocardiogram and nasolaryngoscopy. For the nasolaryngoscopy, the subject's voice box and epiglottis (flap of tissue that covers the windpipe during swallowing) are examined using a thin flexible tube with a camera attached that is passed through the nose to the back of the throat. During the test, speech and other tasks such as singing and whistling are observed. The camera records the movement of the vocal cords on videotape. This procedure may be repeated another time during the study.

Participants undergo the following procedures:

* Electrical stimulation of muscles in the neck: The muscles in the neck are stimulated with brief low-level electrical currents to see if the stimulation can cause the epiglottis to fold down over the windpipe. Stimulation may be increased to a level where it feels like a small shock The subject is asked to try to do the muscle stimulation while swallowing.
* Videofluoroscopy (recording swallowing and muscle stimulation during x-ray imaging of the head): The head and neck are x-rayed while the subject swallows. After the wires have been inserted for EMG (see below), markers are glued to the tongue and a tube is inserted through the nose into the esophagus. The movements during swallowing with and without muscle stimulation are x-rayed and analyzed later to determine how the stimulation affects the movement of the epiglottis.
* Electromyography (EMG): Measurement of the electrical activity of muscles in the neck using fine wires placed through the skin into muscles in the chin.
* Manometry: During the videofluoroscopy, a manometer (tube that measures pressures) is placed through the nose and into the back of the throat at the entry point to the esophagus. This test shows whether muscle stimulation can fold down the epiglottis.
* Surface electromyography (sEMG): The tube used during the videofluoroscopy has small rings embedded in it that measure muscle activity on the surface of the inside of the throat.

DETAILED DESCRIPTION:
OBJECTIVE:

Our objective is to determine the factors that cause epiglottic inversion during normal deglutition and attempt to recreate this movement by means of muscle stimulation.

STUDY POPULATION:

We plan to accrue 30 healthy volunteers so that a set of 20 participants will provide reliable data for analysis.

DESIGN:

As an observational study, anatomical movement will be examined with videofluoroscopy during normal swallows and during stimulation of the thyrohyoid, geniohyoid, hyoglossus, and styloglossus muscles.

OUTCOME MEASURES:

The principal outcome of this study is the distance of epiglottal displacement as measured from videofluoroscopic images during normal swallowing and muscle stimulation. Secondary measures are assessed as correlates of epiglottal inversion. These data include motion and kinematics of other structures, such as the hyo-laryngeal complex and the tongue; tongue base retraction pressures in the oral-pharynx, the hypopharynx, and the UES; and muscle activity as measured by surface electromyography in these three locations.

ELIGIBILITY:
* INCLUSION CRITERIA:

Included subjects will be healthy adults age 18-65 years with normal swallowing function, as determined with a medical history and physical examination by an otolaryngologist.

EXCLUSION CRITERIA:

Exclusion criteria include the following circumstances:

* Subjects must not have a history of chronic swallowing difficulty or dysfunction.
* Pregnant volunteers will be excluded due to risks associated with radiation exposure.
* Women who are nursing will be excluded.
* Subjects must not currently be suffering from a psychiatric disorder other than depression, as evidenced by being under the care of a psychiatrist, or on medications for treatment of a psychiatric disorder.
* History of brain injury or neurological disease.
* History of epileptic seizure.
* History of Rheumatic fever, mitral valve prolapse, heart murmurs, or cardiac arrhythmias as determined by medical history, physical and EKG will disqualify a subject.
* Subjects must not be taking any medications, including herbal types that can affect coagulation.
* Subjects will be excluded if they have a history of allergies to lidocaine or any other anesthetic medication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2007-05-16; Primary Completion 2009-09-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Gresham SL. Clinical assessment and management of swallowing difficulties after stroke. Med J Aust. 1990 Oct 1;153(7):397-9. doi: 10.5694/j.1326-5377.1990.tb125497.x. PMID 2215310
- [Background] DOTY RW, BOSMA JF. An electromyographic analysis of reflex deglutition. J Neurophysiol. 1956 Jan;19(1):44-60. doi: 10.1152/jn.1956.19.1.44. No abstract available. PMID 13286721
- [Background] Logemann JA, Kahrilas PJ, Cheng J, Pauloski BR, Gibbons PJ, Rademaker AW, Lin S. Closure mechanisms of laryngeal vestibule during swallow. Am J Physiol. 1992 Feb;262(2 Pt 1):G338-44. doi: 10.1152/ajpgi.1992.262.2.G338. PMID 1539666